CLINICAL TRIAL: NCT07261306
Title: Comparison Between Oral Methotrexate and Tofacitinib in Chronic Plaque Psoriasis
Acronym: MTX
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Lahore General Hospital (Other Government)
Responsible Party: Principal Investigator, Maryam Fatima, Principal Investigator, Lahore General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Derma LGH
Record Dates: First submitted 2025-07-23; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-08

CONDITIONS: Psoriasis
Keywords: MtX; Tofacitinib
MeSH Terms: conditions — Psoriasis | interventions — Methotrexate; tofacitinib

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group mTX (Active Comparator): Methotrexate is a modified antirheumatic drug work by inhibiting dihydrofolate reductase
  Interventions: Drug: Methotrexate
- Tofacitinib (Active Comparator): Tofacitinib is janus kinase inhibitor and had a role in treatment of psoriasis and psoriatic arthritis
  Interventions: Drug: Tofacitinib

INTERVENTIONS:
Drug: Methotrexate — Methotrexate is an antifolate drug work by inhibiting enzyme dihydrofolate reductase and inhibit cell proliferation and play a role in psoriasis treatment
  Arms: Group mTX
Drug: Tofacitinib — Tofacitinib is janus kinase inhibitor and have role in psoriasis
  Arms: Tofacitinib

SUMMARY:
Psoriasis is a chronic inflammatory dermatoses which include well demarcated scaly erythematous plaques on whole body including scalp role of methotrexate vs tofacitinib is compared in this study

DETAILED DESCRIPTION:
Comparison between safety and efficacy of oral methotrexate and tofacitinib in chronic plaque psoriasis is to be determined in this study

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18- 70 years of either gender.
* Only patients with Psoriasis Area and Severity Index (PASI) score of 10 or above, and/or Body Surface Area (BSA) involvement of 10% or more, will be included.
* Duration of plaque psoriasis for at least 6 months prior to the study.
* Psoriasis that has not shown adequate response to topical therapies

Exclusion Criteria:

* Individuals with other forms of psoriasis or other significant dermatological conditions that might interfere with the assessment of psoriasis.
* Participants currently receiving systemic corticosteroids, biologics, or any other immunosuppressive agents within 4 weeks prior to the start of the study will be excluded.
* Known hypersensitivity or contraindications to either methotrexate or tofacitinib.
* History of significant liver, kidney, hematologic/bleeding disorder, gastrointestinal/acid peptic disease, or immune system disorders.and any history of tuberculosis and malignancy.
* Pregnant or lactating women will not be eligible for the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-08-29 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
Efficacy Achievement | Baseline to Week 12 of treatment
  The primary outcome will be the proportion of participants who demonstrate a minimum 75 percent reduction in the Severity Index (PASI-75) from baseline to Week 12 of treatment. A participant will be classified as "Achieved" if the Week-12 PASI score reflects a reduction of 75 percent or greater from the baseline measurement, and "Not Achieved" if this threshold is not met.

SECONDARY OUTCOMES:
Percentage Reduction in PASI Score | From Baseline to Week 12
  This outcome will quantify the degree of improvement by calculating the percentage reduction in PASI score from baseline to Week 12. Percentage reduction will be computed using the formula:
  [(Baseline PASI - Week-12 PASI) ÷ Baseline PASI] × 100.

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Fatima, Principal Investigator — Lahore General Hospital, Lahore
Locations (1):
- Lahore general hospital, Lahore, Punjab Province, Pakistan